CLINICAL TRIAL: NCT06639451
Title: A Prospective, Multi-center Study to Evaluate Efficacy and Safety of BSJ020R in Treatment of AVF for Hemodialysis
Brief Title: A Prospective, Multi-center Study to Evaluate Efficacy and Safety of BSJ020R in Treatment of AVF for Hemodialysis (RANGER AV Japan Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2511
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Arteriovenous Fistula Stenosis; Arteriovenous Fistula; Vascular Access
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RANGER™ Paclitaxel Coated Balloon (Experimental): RANGER™ Paclitaxel Coated Balloon Catheter angioplasty in the AVF at the index procedure.
  Interventions: Device: RANGER™ Paclitaxel Coated Balloon Catheter

INTERVENTIONS:
Device: RANGER™ Paclitaxel Coated Balloon Catheter — A procedure that utilizes a balloon coated with paclitaxel (drug) which can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a balloon coated with paclitaxel at the end of it. When the tube is in place, it inflates to open the blood vessel, so that normal blood flow is restored. The tube is then removed.

SUMMARY:
A prospective, multi-center study to evaluate efficacy and safety of BSJ020R in treatment of AVF for hemodialysis

DETAILED DESCRIPTION:
Primary objective of this study is to evaluate the effectiveness and safety of the Ranger™ Paclitaxel Coated Balloon Catheter for treating subjects presenting with de novo or non-stented restenotic lesions of native arteriovenous dialysis fistulae (AVF) in the upper extremity.

The primary endpoint is the target lesion primary patency (TLPP) rate at 6 months post index procedure. Primary patency is a binary endpoint, defined as freedom from clinically-driven target lesion revascularization (clinically-driven TLR) or access circuit thrombosis measured at 6 months post index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide consent before any study-specific tests or procedures are performed and agree to attend all required follow-up visits.
2. Subject at least 18 years of age.
3. Subject has a native AV fistula created ≥ 60 days prior to enrollment.
4. The target AVF has undergone successful dialysis for at least 8 of 12 sessions during a four-week period prior to enrollment.
5. Subjects on stable dialysis has all of the following criteria meet.

   * No significant decrease in blood pressure during dialysis during a four-week period prior to enrollment
   * No significant edema
   * No signs of heart failure
6. Target lesion is located between the arteriovenous anastomosis and axillosubclavian junction.

   Note: If the lesion is in the anastomosis, the treatment may be delivered up to 2 cm upstream on the arterial side. Note: If the lesion is in the cephalic arch, the treatment may be delivered up to 2 cm into the subclavian vein.
7. Angiographic evidence that target lesion consists of a de novo and/or non-stented restenotic lesion with ≥ 50% stenosis by visual estimate.
8. Most recent standard PTA (ie. non-drug coated) treatment must be > 3 months prior to enrollment and most recent DCB treatment must be > 6 months prior to enrollment.
9. A target lesion with total lesion length up to 130 mm by visual estimate. Note: Tandem (or "adjacent") lesions may be enrolled provided they meet all of the following criteria:

   1. Separated by a gap of ≤ 30mm (3 cm).
   2. Total combined lesion length, including 30 mm gap, is ≤ 130 mm.
   3. Able to be treated as a single lesion.
10. Reference vessel diameter ≥ 4.0 mm and ≤ 8.0 mm by visual estimate.
11. Subject underwent successful crossing of the target lesion with the guide wire and pre-dilatation with only high pressure PTA balloon(s) defined as:

    1. Residual stenosis of ≤ 30% AND.
    2. Absence of a flow limiting dissection (Grade ≥ C) or perforation.

Exclusion Criteria:

1. Life expectancy, documented in the investigator's opinion, of less than 12 months.
2. Receiving immunosuppressive therapy.
3. Anticipating a kidney transplant within 6 months of enrollment into the study.
4. Patient with anticipated conversion to peritoneal dialysis.
5. Patient with AVF infection or systemic infection.
6. Patient has planned surgical revision of AVF.
7. Presence of secondary non-target lesion requiring treatment within 30-days post index procedure.
8. Patient with hemodynamically significant central venous stenoses that cannot be successfully treated prior to treatment of the target lesion.
9. Patient with target AVF or access circuit which had within 1 year prior to enrollment or currently has a thrombosis.
10. Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon or proper placement of the delivery system.
11. Target lesion located central to the axillosubclavian junction.
12. Patient has significant arterial inflow lesion requiring treatment more than 2 cm upstream from the anastomosis in the AVF.
13. Presence of aneurysm requiring treatment at the lesion site.
14. Presence of a stent or graft located in the target access circuit.
15. Known allergies or sensitivities to paclitaxel and/or raw materials of test devices including ATBC (refer to Kiki-gaiyosho).
16. Known contraindication, including allergic reaction, or sensitivity to contrast material that, in the opinion of the investigator, cannot be adequately pretreated.
17. Patient who cannot receive antiplatelet and/or anticoagulant therapy in accordance with the investigator's direction.
18. Clinically significant Steal Syndrome requiring treatment.
19. Women who are breastfeeding, pregnant, or the subject with known intention to procreate within 6 months after index procedure. Note: 6-month contraception after index procedure is required.
20. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint, or subject was previously enrolled in this study.
21. Subject intends to participate in another investigational drug or device clinical trial within 6 months after the index procedure.
22. Patient has a co-morbid condition that, in the opinion of the investigator, may cause him/her to be non-compliant with the protocol or confound the data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion primary patency rate | 6 months post index procedure
  Primary patency is a binary endpoint, defined as freedom from clinically-driven target lesion revascularization (clinically-driven TLR) or access circuit thrombosis measured at 6 months post index procedure.
  Note: Clinically-driven TLR is defined as any re-intervention involving the target lesion in which:
  * The subject has a ≥50% diameter stenosis (per angiographic core laboratory assessment) in the presence of clinical or physiologic abnormalities that indicate dialysis access dysfunction OR
  * ≥70% stenosis (per angiographic core laboratory assessment) without the presence of clinical or physiologic abnormalities indicating dialysis access dysfunction

OTHER OUTCOMES:
Technical success | Day of index procedure
  Technical success defined as successful delivery, inflation, deflation and retrieval of the intact study balloon device without burst at or below rated burst pressure (RBP)
Procedure success | Day of index procedure
  Procedure success defined at maintenance of patency (≤30% residual stenosis) confirmed by the core laboratory in the absence of serious adverse device effect (SADE) on the day of index procedure.
Clinical success | 12 months post-index procedure
  Clinical success defined as resumption of successful dialysis for at least one session after index procedure and before re-intervention.
Access circuit primary patency | 3, 6, 9 and 12 months post-index procedure
  Access circuit primary patency defined as freedom from re-intervention in the access circuit or access circuit thrombosis.
Target lesion primary patency | 3, 9 and 12 months post-index procedure
  Target lesion primary patency defined as freedom from clinically-driven TLR or access circuit thrombosis occurring in the target lesion.
Rate of clinically-driven TLR and TLR | 3, 6, 9 and 12 months post-index procedure
Rate of intervention required to maintain access circuit patency | 3, 6, 9 and 12 months post-index procedure
  Rate of intervention required to maintain access circuit patency defined as re-interventions in the target lesion and/or access circuit through 12 months.
Serious Adverse Events (SAEs) involving the AV Access circuit | 1, 3, 6, 9 and 12 months post-index procedure
Device related adverse event rate | 1, 3, 6, 9, and 12 months post-index procedure
Procedure related adverse events rate | 12 months post-index procedure
Quality of Life | 3, 6, and 12 months post-index procedure
  Quality of Life assessed by EuroQol 5 dimensions (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Tomonari Ogawa, MD, Principal Investigator — Saitama Medical Center
Locations (8):
- Japan (8):
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Yokohama Dai-ichi Hospital, Yokohama, Kanagawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Osaka Keisatsu Hospital, Osaka, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Shizuoka General Hospital, Shizuoka, Shizuoka
  - Saiseikai Central Hospital, Minato, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama

IPD SHARING:
Plan to Share IPD: No
No plan so far, but the anonymized data and study protocol for this clinical trial may be made available to other researchers in accordance with Boston Scientific Data Sharing Policy: (http://www.bostonscientific.com/en-US/data-sharing-requests.html)